CLINICAL TRIAL: NCT00584246
Title: Pregabalin (Lyrica) for the Treatment of Restless Legs Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to budget (personnel) limitations.
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Theresa Zesiewicz, MD, Professor of Neurology, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3; 105362
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome; RLS; Pregabalin; Lyrica
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pregabalin (Lyrica)
  Interventions: Drug: Pregabalin (Lyrica)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Pregabalin (Lyrica); Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin (Lyrica) — 50 - 150 mg po qhs for 2 months
Drug: Placebo — 50 - 150 mg po qhs for 2 months
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of Pregabalin (Lyrica) in treating patients with Restless Legs Syndrome (RLS) in a double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with RLS diagnosed by a movement disorder specialist/ Sleep specialist .
2. Patients must report some degree of pain which occurs on a regular basis.
3. Age 18 years to 80 years.
4. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
5. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
6. Willing and able to provide informed consent.
7. Willing to comply with protocol. -

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study.
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Current treatment with a dopamine agonist (unless stopped at least 2 weeks prior to baseline).
5. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 24).
6. Legal incapacity or limited legal capacity.
7. Presence of severe renal disease BUN 50% greater than normal, Patients must have evidence from their PCP or Urologists of normal PSA and urodynamic tests within the last 12 month. Normal BUN levels should be within a range of 5 to 20 mg/ d L and creatinine between .7 and 1.4 mg/ d L. Labs will be requested from PCP.
8. Presence of major hepatic impairment (Cirrhosis, Viral Hepatitis, Nonalcoholic Steatohepatitis, Wilson's disease, or Hemochromatosis). LFT must show non-clinically significant results (Albumin range 3.0-6.0; Alkaline phosphatase range 40-150; ALT range 0-55; AST range 5-34).
9. Presence of severe daytime sleepiness.
10. Present complaints of somnolence, dizziness, blurred vision, bleeding tendencies, cardiac abnormalities.
11. Patients taking dopamine agonists for any condition other than RLS. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
International RLS Study Group Severity Scale (IRLS) | 2 months

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States